CLINICAL TRIAL: NCT04254978
Title: A Phase 2 Multi-Center, Open Label Study to Assess the Safety, Efficacy and Pharmacodynamics of IMG-7289 in Patients With Essential Thrombocythemia
Brief Title: Study of Bomedemstat in Participants With Essential Thrombocythemia (IMG-7289-CTP-201/MK-3543-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imago BioSciences, Inc., a subsidiary of Merck & Co., Inc., (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMG-7289-CTP-201; MK-3543-003 (Other: Merck); 2019-003659-13 (EudraCT Number)
Record Dates: First submitted 2020-01-15; First posted 2020-02-05 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Essential Thrombocythemia
MeSH Terms: conditions — Thrombocythemia, Essential | interventions — bomedemstat

STUDY DESIGN:
Intervention Model Description: Multi-center, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bomedemstat (Experimental): Bomedemstat administered daily for 169 consecutive days
  Interventions: Drug: Bomedemstat

INTERVENTIONS:
Drug: Bomedemstat — Oral administration
  Other Names: IMG-7289; MK-3543

SUMMARY:
This is a Phase 2b open label study of an orally administered LSD1 inhibitor, Bomedemstat (MK-3543, formerly called IMG-7289), in patients with essential thrombocythemia.

This study investigates the following:

* The safety and tolerability of Bomedemstat
* The pharmacodynamic effect of Bomedemstat

DETAILED DESCRIPTION:
This is a Phase 2 multi-center, open-label study evaluating the safety, efficacy and pharmacodynamics of Bomedemstat administered orally once daily in patients with essential thrombocythemia (ET). Patients will be dosed with Bomedemstat for 169 consecutive days in the Initial Treatment Period (ITP). Qualifying patients may continue to receive Bomedemstat in the Additional Treatment Period (ATP).

Safety will be evaluated by clinical assessments of safety parameters i.e., safety laboratory testing, adverse event reporting, physical examination and vital sign assessments. Pharmacodynamics will be evaluated by hematology assessment, patient reported symptom burden, change in spleen size by palpation and other measures.

To ensure safety, a Safety Advisory Board will perform periodic reviews of safety parameters and pharmacodynamic markers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Essential Thrombocythemia per World Health Organization (WHO) diagnostic criteria for myeloproliferative neoplasms.
* Requires treatment in order to lower platelet count based on patient age over 60 or history of thrombosis.
* Have failed at least one standard therapy
* Must have discontinued ET therapy at least 1 week (4 weeks for interferon) prior to study drug initiation.

Exclusion Criteria:

* Has undergone major surgery ≤4 weeks prior to starting study drug or has not recovered from side effects of such surgery.
* Unresolved treatment related toxicities from prior therapies (unless resolved to ≤ Grade 1).
* Uncontrolled active infection.
* Current use of prohibited medications
* Known HIV infection or active Hepatitis B or Hepatitis C virus infection
* Other hematologic/biochemistry requirements, as per protocol
* Use of investigational agent within last 14 days
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (25):
- United States (7):
  - Local Institution, Jacksonville, Florida
  - Local Institution, Ann Arbor, Michigan
  - Local Institution, New York, New York
  - Local Institution, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Seattle, Washington
- Australia (6):
  - Local Institution, Herston, Brisbane
  - Local Institution, Camperdown, New South Wales
  - Local Institution, St Leonards, New South Wales
  - Local Institution, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Local Institution, Clayton, Victoria
- Germany (2):
  - Department of Hematology and Stem Cell Transplantation, West German Cancer Center (WTZ), Essen
  - Local Institution, Jena
- Local Institution, Hong Kong, Hong Kong
- Italy (4):
  - Local Institution, Alessandria
  - Local Institution, Bologna
  - CRIMM; Centro Ricerca e Innovazione delle Malattia Mieloproliferative, Azienda ospedaliera Universitaria Careggi, Florence
  - Local Institution, Varese
- New Zealand (2):
  - Local Institution, Auckland
  - Middlemore Hospital, Auckland
- United Kingdom (3):
  - Local Institution, London
  - Guys and St Thomas Hospital, London
  - Local Institution, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Bomedemstat: Bomedemstat was administered daily for 169 consecutive days of the initial treatment period. After completing 169 days of treatment, qualifying participants continued into additional treatment periods of 169 days each, for as long as the participant continued to derive clinical benefit.
Period: Initial Treatment Period (ITP)
Arm/Group | Bomedemstat
Started | 73
Completed | 64
Not Completed | 9
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 1
Period: Additional Treatment Period (ATP)
Arm/Group | Bomedemstat
Started | 63 (One participant completed the ITP but did not continue into the additional treatment period)
Completed | 52
Not Completed | 11
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Arm/Group | Bomedemstat
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.8 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 51
  More than one race | 0
  Unknown or not reported | 0
  Aboriginal | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any undesirable physical, psychological or behavioral effect experienced by a participant during the study, in conjunction with the use of the drug or biologic, whether or not product related. This includes any untoward signs or symptoms experienced by the participant from the time of first dose with study treatment until completion of the study. The number of participants who experienced an AE is reported.
Time Frame: Up to approximately 30 months
Population: All participants who were enrolled in the study and received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Bomedemstat: Bomedemstat was administered daily for 169 consecutive days of the initial treatment period. After completing 169 days of treatment, qualifying patients continued into additional treatment periods of 169 days each, as long as the participant continued to derive clinical benefit.
Arm/Group | Bomedemstat
Number analyzed (Participants) | 73
Participants | 73

2. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is any undesirable physical, psychological or behavioral effect experienced by a patient during participation in the study, in conjunction with the use of the drug or biologic, whether or not product-related. This includes any untoward signs or symptoms experienced by the patient from the time of first dose with study treatment until completion of the study. The number of participants who discontinued study treatment due to an AE is reported.
Time Frame: Up to approximately 28 months
Population: All participants who were enrolled in the study and received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Bomedemstat
Number analyzed (Participants) | 73
Participants | 11

3. Primary Outcome: Percentage of Participants With Platelet Count ≤400 k/μL at Day 169
Description: Blood samples were collected at pre-specified timepoints to determine platelet counts. The percentage of participants who achieved reduction in platelet count to ≤400k/μL in the absence of new thrombolytic events is reported.
Time Frame: Up to day 169
Population: All participants who were enrolled in the study, received at least one dose of study drug, and had a non-missing baseline and at least 1 non-missing post-baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Bomedemstat: Bomedemstat was administered daily for 169 consecutive days
Arm/Group | Bomedemstat
Number analyzed (Participants) | 64
Percentage of Participants | 76.6 [64.3 to 86.2]
Statistical Analysis 1: Comparison: Bomedemstat; Comparison of the true response rate of bomedemstat to a fixed efficacy target of 5%: Null hypothesis (H0): p ≤ 0.05 versus alternate hypothesis (H1): p > 0.05; Test type: Superiority; p < .0001, Exact binomial distribution

ADVERSE EVENTS:
Time Frame: Up to approximately 30 months
Description: The all cause mortality population includes all participants enrolled and randomized in the study. The serious adverse event (AE) and other AE population includes all participants who were enrolled in the study and received at least one dose of study drug.
Arm/Group | Bomedemstat
All-Cause Mortality (participants affected / at risk) | 2/73
Serious Adverse Events (participants affected / at risk) | 27/73
Other Adverse Events (participants affected / at risk) | 72/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bomedemstat (N=73)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Ileal ulcer (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Rotator cuff repair (Surgical and medical procedures) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bomedemstat (N=73)
Anaemia (Blood and lymphatic system disorders) | 14 (35)
Neutropenia (Blood and lymphatic system disorders) | 8 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 23 (47)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 29 (35)
Diarrhoea (Gastrointestinal disorders) | 15 (22)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Flatulence (Gastrointestinal disorders) | 4 (4)
Gingival bleeding (Gastrointestinal disorders) | 6 (6)
Haemorrhoids (Gastrointestinal disorders) | 4 (4)
Large intestine polyp (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 10 (17)
Vomiting (Gastrointestinal disorders) | 5 (5)
Fatigue (General disorders) | 21 (35) — General disorders and administration site conditions
Influenza like illness (General disorders) | 9 (10) — General disorders and administration site conditions
Oedema peripheral (General disorders) | 11 (15) — General disorders and administration site conditions
COVID-19 (Infections and infestations) | 19 (19)
Cellulitis (Infections and infestations) | 4 (5)
Gastroenteritis (Infections and infestations) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 4 (6)
Urinary tract infection (Infections and infestations) | 5 (9)
Contusion (Injury, poisoning and procedural complications) | 18 (25)
Limb injury (Injury, poisoning and procedural complications) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4)
Blood creatinine increased (Investigations) | 4 (8)
Weight decreased (Investigations) | 7 (8)
Decreased appetite (Metabolism and nutrition disorders) | 6 (8)
Gout (Metabolism and nutrition disorders) | 4 (5)
Iron deficiency (Metabolism and nutrition disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (75)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (9)
Joint effusion (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (18)
Dizziness (Nervous system disorders) | 11 (12)
Dysgeusia (Nervous system disorders) | 43 (62)
Headache (Nervous system disorders) | 12 (26)
Paraesthesia (Nervous system disorders) | 5 (10)
Syncope (Nervous system disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 6 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (17)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (17)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (4)
Hot flush (Vascular disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Lead/Coordinating Investigator will have the right to submit for publication any results arising from the study subject to the terms and conditions of the Clinical Trial and Confidentiality Disclosure Agreements.

DOCUMENTS (2):
  • Study Protocol (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT04254978/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT04254978/SAP_001.pdf